CLINICAL TRIAL: NCT05144022
Title: Multi-level Molecular Profiling of High Acute Stress
Brief Title: Multi-level Molecular Profiling of High Acute Stress: a Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Dr. Nils Gassen, Principal Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HighStress
Record Dates: First submitted 2021-10-27; First posted 2021-12-03 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Stress; Bungee Jump; Autophagy

STUDY DESIGN:
Intervention Model Description: 2 groups each undergoing one out of two conditions ("high stress" (bungee jump) or "no stress" (control))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventions group: High stress condition (bungee jump) (Experimental): 25-30 healthy male volunteers participating in a bungee jump
  Interventions: Behavioral: Bungee jump
- Control group: No stress condition (Placebo Comparator): 10-15 healthy males serving as a control group without undergoing a stress event/intervention
  Interventions: Behavioral: Bungee jump

INTERVENTIONS:
Behavioral: Bungee jump — Bungee jump from a cran

SUMMARY:
Although it is well known that stress plays an important role in the development of neuropsychiatric diseases, the precise role and molecular effects of stress have only been poorly understood. For example, autophagy is essential for energy and cellular homeostasis through protein catabolism, and dysregulation results in compromised proteostasis, stress-coping behavior, and excessive secretion of signaling molecules and inflammatory factors. Therefore, the aim of the project is to analyze the clinical effects of a bungee jump resembling an acute stress event in correlation to autophagy and other underlying, multi-level molecular profiling. Specifically, it is planned to perform multi-level molecular profiling and sleep analysis in a cohort of healthy male individuals before, during, and after a bungee jump compared to a control cohort of healthy males not undergoing a stress event. The resulting findings will advance the role of autophagy during the stress response and hence in the development of psychiatric disorders, and possibly investigate alternative treatment venues on a molecular level, and finally contribute to a better clinical outcome.

DETAILED DESCRIPTION:
Although it is well known that stress plays an important role in the development of neuropsychiatric diseases, the molecular effects of stress have only been poorly understood. So far it is known that stress leads to an activation of the stress hormone axis followed by an increased release of the stress hormone and glucocorticoid cortisol. Glucocorticoids bind to glucocorticoid receptors that initiate a cellular signal cascade. However, it can be assumed that other factors are involved but a profound understanding of the stress response at the molecular level has not yet been performed yet.

Using a so-called "multi-omics approach" it is possible to determine changes in a large number of molecular groups, such as proteins or lipids to research the underlying mechanisms of diseases. While multi-omics analyzes have already helped gain elementary knowledge in a large number of somatic diseases, the molecular effects of acute stress have not been addressed yet. This will be the primary focus of this study. To achieve this an acute, concise stress reaction closely resembling a genuine stress response is desired. In previous studies, it was shown that bungee jumping triggers such a short, intense stress reaction and the corresponding activation of the stress hormone axis.

To achieve this a cohort of 25-30 healthy male individuals who undergo a bungee jump resembling an acute stress event will be compared to a cohort of 10-20 healthy males who undergo the same experimental design without undertaking a bungee jump or other stress intervention. At different time points (baseline, shortly before and after the intervention, at multiple time points during the intervention as well as around one week follow up after the intervention) serval psychometrical questionnaires will be gathered and blood will be collected. A dexamethasone inhibition test will be performed before the stress intervention. Sleep quality will be additionally assessed during the entire course of the study by actigraphy. On selected days blood will be collected. Following, autophagy activity will be assessed by Western Blot analysis, and mass spectrometry-based proteomics, phosphoproteomics, metabolomics, and lipidomics will be performed. Bioinformatic analysis, statistical evaluation, quality control, and in silico pathway analyses will then specifically identify factors and cascades of relevance.

The aim of the project is to analyze the clinical effects of an acute stress event in correlation to the underlying, multi-level molecular profiling. Longitudinal multi-omic profiling including proteome, metabolome, lipidome, and epigenetic changes will reveal time-series analysis of thousands of molecular changes and an orchestrated composition of autophagy depended signaling. The resulting findings will advance the role of autophagy in the development of psychiatric disorders, and possibly investigate alternative treatment venues on a molecular level, and finally contribute to a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Present written declaration of consent
* Healthy
* Male
* BMI between 18,5 and 24,9 and body weight between 50kg and 120kg

Exclusion Criteria:

* Insufficient linguistic communication
* Drug abuse or alcohol dependency
* regular medication except for L-thyroxine or antihistamines
* known severe eye disease or severely impaired eyesight or hearing
* a known disease of the cardiovascular system, hypertension higher than 160/90mmHg
* known pulmonary disease, e.g. bronchial asthma
* known fractures of the spine or skeletal system of the lower extremity
* surgery within the last 4 to six months
* intervention group: fear of heights

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Proteomics and autophagy processes | change from baseline to the stress intervention and a 5- 7 day follow up
  Change in protein levels of autophagy biomarkers (LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting.

SECONDARY OUTCOMES:
Proteome patterns | change from baseline to the stress intervention and a 5- 7 day follow up
  Change in protein levels and protein phosphorylation by untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells).
Metabolic processes | change from baseline to the stress intervention and a 5- 7 day follow up
  Metabolic measurements by mass spectrometry, in order to determine variations in plasma metabolites, including targeted analysis of steroid hormones
Lipid profiling | change from baseline to the stress intervention and a 5- 7 day follow up
  Targeted and quantitative analysis by mass spectrometry of change in plasma Lipids.
Saliva Cortisol Levels | comparison between groups
  Saliva Cortisol Levels in nmol per Liter (nmol/L) after dexamethasone intake will be evaluated and compared ton the control group
Sleep Efficiency | change from baseline to the stress intervention and a 5- 7 day follow up
  Assessment of Sleep Efficiency (total time in bed/time asleep during night) by GenActive Actigraphs
Overall sleep Quality | change from baseline to the stress intervention and a 5- 7 day follow up
  Sleep diary to assess overall sleep quality assessed as ratio of the total time spent asleep (in hours) to the total amount of time spent in bed (in hours) per night
Sleep Quality (PSQI) | change from baseline to the stress intervention and a 5- 7 day follow up
  Pittsburgh Sleep Quality Index (PSQI): self-report questionnaire to assess sleep quality over a 1-month time interval consisting of 19 individual items.
Mental well-being (WEMWBS) | change from baseline to the stress intervention and a5- 7 day follow up
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS): self-reported 14-item scale to assess Overall mental wellbeing, minimum value 14, maximum value 70, high score indicating high well-being
Resilience behavior (Wagnild &Young) | change from baseline to the stress intervention and a 5- 7 day follow up
  Resilience scale (Wagnild &Young): self-reported 25-item scale to assess overall resilience, minimum value 25, maximum value 175, high score indicating higher resilience
Phosphoproteome patterns | change from baseline to the stress intervention and a 5- 7 day follow up
  Change in protein phosphorylation by untargeted mass spectrometry-based phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells).
Ubiquitinome patterns | change from baseline to the stress intervention and a 5- 7 day follow up
  Change in protein ubiquitination levels by untargeted mass spectrometry-based proteomics of isolated PBMCs (peripheral blood mononuclear cells).

CONTACTS AND LOCATIONS:
Overall Officials: Nils Gassen, Dr. rer. nat., Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Clinic for psychiatry and psychotherapy, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayash S, Schmitt U, Lyons DM, Muller MB. Stress inoculation in mice induces global resilience. Transl Psychiatry. 2020 Jun 19;10(1):200. doi: 10.1038/s41398-020-00889-0. PMID 32561821
- [Background] Hasin Y, Seldin M, Lusis A. Multi-omics approaches to disease. Genome Biol. 2017 May 5;18(1):83. doi: 10.1186/s13059-017-1215-1. PMID 28476144
- [Background] Hennig J, Laschefski U, Opper C. Biopsychological changes after bungee jumping: beta-endorphin immunoreactivity as a mediator of euphoria? Neuropsychobiology. 1994;29(1):28-32. doi: 10.1159/000119059. PMID 8127421
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] de Kloet ER, Joels M, Holsboer F. Stress and the brain: from adaptation to disease. Nat Rev Neurosci. 2005 Jun;6(6):463-75. doi: 10.1038/nrn1683. PMID 15891777
- [Background] Leistner C, Menke A. How to measure glucocorticoid receptor's sensitivity in patients with stress-related psychiatric disorders. Psychoneuroendocrinology. 2018 May;91:235-260. doi: 10.1016/j.psyneuen.2018.01.023. Epub 2018 Feb 2. PMID 29449045
- [Background] Lyons DM, Parker KJ, Katz M, Schatzberg AF. Developmental cascades linking stress inoculation, arousal regulation, and resilience. Front Behav Neurosci. 2009 Sep 18;3:32. doi: 10.3389/neuro.08.032.2009. eCollection 2009. PMID 19826626
- [Background] Nicora G, Vitali F, Dagliati A, Geifman N, Bellazzi R. Integrated Multi-Omics Analyses in Oncology: A Review of Machine Learning Methods and Tools. Front Oncol. 2020 Jun 30;10:1030. doi: 10.3389/fonc.2020.01030. eCollection 2020. PMID 32695678
- [Background] van Westerloo DJ, Choi G, Lowenberg EC, Truijen J, de Vos AF, Endert E, Meijers JC, Zhou L, Pereira MP, Queiroz KC, Diks SH, Levi M, Peppelenbosch MP, van der Poll T. Acute stress elicited by bungee jumping suppresses human innate immunity. Mol Med. 2011 Mar-Apr;17(3-4):180-8. doi: 10.2119/molmed.2010.00204. Epub 2010 Dec 10. PMID 21203694